CLINICAL TRIAL: NCT05188872
Title: 68Ga-Pentixafor PET/CT in the Diagnosis of Primary Aldosteronism and Pre-postoperative of Superselective Adrenal Artery Embolization
Brief Title: Application of 68Ga-Pentixafor PET/CT in Primary Aldosteronism and Pre-postoperative of SAAE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director, Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian12
Record Dates: First submitted 2021-08-30; First posted 2022-01-12 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Positron-Emission Tomography
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-Pentixafor (Experimental): Each subject receive a single intravenous injection of 68Ga-Pentixafor, and undergo PET/CT imaging within the specificed time
  Interventions: Diagnostic Test: 68Ga-Pentixafor

INTERVENTIONS:
Diagnostic Test: 68Ga-Pentixafor — Each patient receive a single intravenous injection of 68Ga-Pentixafor, and undergo PET/CT scan within specified time.
  Other Names: PET/CT scan

SUMMARY:
Primary aldosteronism is the most common cause of secondary hypertension. The two main types of primary aldosteronism are aldosteronoma(30%) and adrenal hyperplasia(60%). The gold standard that determines the diagnosis and treatment strategy of primary aldosteronism is adrenal vein sampling(AVS), but the success rate is only about 80%. Using CXCR4 as a probe for 68Ga-Pentixafor PET/CT imaging can guide the classification diagnosis and treatment strategy of primary aldosteronism, which is a favorable supplement to AVS. Superselective adrenal artery embolization(SAAE) and laparoscopy are the main operation treatments for primary aldosteronism. SAAE is an invasive interventional operation. It is a novel way to evaluate the changes in the structure and function of adrenal tissue pre-postoperative SAAE by using the changes in 68Ga-Pentixafor PET/CT imaging.

DETAILED DESCRIPTION:
Primary aldosteronism: Hypertension is divided into primary hypertension and secondary hypertension. Secondary hypertension refers to hypertension with clear etiology. When the etiology is identified and effectively removed or controlled, hypertension as a secondary symptom can be cured or significantly relieved. The most common secondary hypertension is primary aldosteronism. Primary aldosteronism is due to excessive aldosterone secretion in the adrenal cortex, characterized by clinical syndromes of hyperaldosteronism, low renin activity, hypertension and hypokalemia. Compared with essential hypertension, the risk of cardiovascular and cerebrovascular events and the risk of target organ damage in patients with primary aldosteronism were significantly increased. On the contrary, early detection and treatment mean better blood pressure control, lighter target organ damage and better clinical outcomes. The two main types of primary aldosteronism are aldosteronoma(30%) and adrenal hyperplasia(60%). The gold standard that determines the diagnosis and treatment strategy of primary aldosteronism is adrenal vein sampling (AVS), but the success rate is only about 80 %. Therefore, it is necessary to explore a non-invasive examination method as a beneficial supplement to AVS.

ELIGIBILITY:
Inclusion Criteria:

* adult population (aged 18 years or order);
* patients with suspected or new diagnosed Primary aldosteronism (supporting evidence may include MRI, CT, laboratory tests);
* patients who had scheduled 68Ga-BNU-PSMA PET/CT scan;
* patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee;
* healthy volunteers(aged 18 years or order).

Exclusion Criteria:

* patients with pregnancy;
* the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | through study completion,an average of 3 years
  Standardized uptake value (SUV) of 68Ga-Pentixafor for each target or suspected lesion of subject.

SECONDARY OUTCOMES:
SAAE treatment evaluation | through study completion,an average of 3 years
  68Ga-Pentixafor PET/CT imaging to evaluate the changes in the structure and function of adrenal tissue pre-postoperative SAAE.

CONTACTS AND LOCATIONS:
Overall Officials: Liangdi Xie, MD, Study Chair — the First Affiliated Hospital, Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fang Z, Cai H, Zhang Q, Gong J, Zhou W, Xie L, Peng F. Comparative Analysis of Single-Path and Multipath Adrenal Venous Sampling in Primary Aldosteronism. J Interv Cardiol. 2023 Aug 12;2023:8670365. doi: 10.1155/2023/8670365. eCollection 2023. PMID 37601238